CLINICAL TRIAL: NCT05531825
Title: Clinical Evaluation Study of a Device for Detecting Arteriovenous Fistula Vascular Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ai Peng (Other)
Responsible Party: Sponsor-Investigator, Ai Peng, Director of the Department of Nephrology, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: SHSY-IEC-5.0/22K54/P01
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Arteriovenous Fistula Flow Monitoring; Early Detection of Complications of Arteriovenous Fistula; Voiceprint

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal control group: Patients with no disease in the main organs, with well-developed body shape, and with good physiological functions, physical activity abilities and labor abilities.
  Interventions: Device: A device for detecting arteriovenous fistula vascular function
- Newly established arteriovenous fistula group: Chronic kidney disease stage 5 (CKD5) non-dialysis patients planning to undergo internal arteriovenous fistula surgery.
  Interventions: Device: A device for detecting arteriovenous fistula vascular function
- reconstructed arteriovenous fistula group: Patients with maintenance hemodialysis who need to reconstruct the internal arteriovenous fistula on account of dissatisfaction with blood flow.
  Interventions: Device: A device for detecting arteriovenous fistula vascular function
- Long-term maintenance hemodialysis group: Patients undergoing hemodialysis with long-term fixed internal arteriovenous fistula.
  Interventions: Device: A device for detecting arteriovenous fistula vascular function

INTERVENTIONS:
Device: A device for detecting arteriovenous fistula vascular function — An innovative design based on PVDF piezoelectric membrane by combining all kinds of technologies including NB-iot/4G transmission mode to realize real-time monitoring and feedback of the health status of arteriovenous fistula vessels

SUMMARY:
Evaluation on the reliability, practicability and safety of a wearable device for measuring arteriovenous fistula function based on voice print.

DETAILED DESCRIPTION:
Arteriovenous fistula is the lifeline of maintenance hemodialysis patients. At present, there is a lack of a simple wearable real-time evaluation technology and device for arteriovenous fistula, which can help doctors find and deal with the complications of arteriovenous fistula timely and accurately. This study proposes an innovative design based on PVDF piezoelectric membrane by combining all kinds of technologies including NB-iot/4G transmission mode to realize real-time monitoring and feedback of the health status of arteriovenous fistula vessels, so that the use time of arteriovenous fistula can be prolonged and the survival rate of dialysis patients can also be improved.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75.
* Patients diagnosed with end-stage renal failure and planning to undergo venous fistula surgery or maintenance hemodialysis.
* Sign the informed consent.

Exclusion Criteria:

* Pregnant and lactating women, bipolar disorder, schizophrenia and other serious mental illness.
* Other circumstances deemed inappropriate by the researcher
* Quit midway

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage renal disease undergoing or planning regular hemodialysis with autologous arteriovenous fistulas
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between voiceprint spectrum and the blood flow of arteriovenous fistula | 2 month
  Correlation between voiceprint spectrum and the blood flow of arteriovenous fistula

CONTACTS AND LOCATIONS:
Overall Officials: Ai Peng, MD,PhD, Study Director — Shanghai 10th People's Hospital
Locations (1):
- Department of Nephrology & Rheumatology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No